CLINICAL TRIAL: NCT00292058
Title: Comparing Patient Outcomes and Cost of Psychiatric Care Provided Through Videoconferencing With Psychiatric Care Provided In-person.
Brief Title: Comparing Telepsychiatry and In-person Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Collaborators: Ontario Mental Health Foundation (Other Government); NORTH Network (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 07911E; 7764101; R2354A01
Record Dates: First submitted 2006-02-14; First posted 2006-02-15 (Estimated); Last update posted 2019-09-25 (Actual); Status verified 2006-02

CONDITIONS: Psychiatric Disorders
Keywords: Telepsychiatry; Videoconference; Psychiatric consultation; Equivalence trial
MeSH Terms: conditions — Mental Disorders

INTERVENTIONS:
Device: Videoconference equipment (telepsychiatry)

SUMMARY:
Psychiatric consultation and short-term follow-up will produce equivalent clinical outcomes and be less costly when provided via videoconferencing (telepsychiatry) than when provided in-person.

DETAILED DESCRIPTION:
We predict that patients referred by their family physician for a psychiatric consultation and, if needed, short-term follow-up will have equivalent clinical outcomes when seen via telepsychiatry as compared to those patients seen in-person. We also predicted that telepsychiatry will be cheaper than in-person care.Study Design: a single-centre equivalence trial.We will use a sample size calculation and analytical methods that are specifically tailored for equivalence trials.

ELIGIBILITY:
Inclusion Criteria:

* patients referred by their family physicians for psychiatric consultation
* scores in the dysfunctional range on the Brief Symptom Inventory

Exclusion Criteria:

* patients incapable of consenting to the research
* patients referred for medico-legal or insurance reports

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495
Dates: Start 2001-08; Study Completion 2004-08

PRIMARY OUTCOMES:
Brief Symptom Inventory
Cost of providing the psychiatric services

SECONDARY OUTCOMES:
Quality of Life Inventory
Client Satisfaction Questionnaire
Hospital Utilization

CONTACTS AND LOCATIONS:
Overall Officials: Richard L O'Reilly, M.B., Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario, Canada